CLINICAL TRIAL: NCT05757765
Title: Medication (de)Prescribing in Hospitalized Geriatric Patients With Sarcopenia, Less is More
Brief Title: (De)Prescribing in Hospitalized Sarcopenic Geriatric Patients
Acronym: MEDEGESARC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZuyderlandMC
Record Dates: First submitted 2023-02-23; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Sarcopenia
Keywords: Polypharmacy; Deprescribing; Geriatric patients
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- deprescribing pharmacotherapy approach (DPA) (Experimental): A new way of medication review in patients with sarcopenia. This method is based on previous scientific research and is aimed at minimizing pharmacotherapy. The aim is to combat symptoms and complaints and to stop (preventive) medication as much as possible
  Interventions: Other: deprescribing pharmacotherapy approach (DPA)
- STOPP-START deprescribing approach (SSA) (Active Comparator): The usual care in the geriatric medicine in the Netherlands consisting of a medication review based on the STOPP-START criteria. These criteria have been combined in a protocol that describes when certain medication(groups) must be continued or discontinued for specific patient characteristics.
  Interventions: Other: STOPP-START deprescribing approach (SSA)

INTERVENTIONS:
Other: deprescribing pharmacotherapy approach (DPA) — A new way of medication review in patients with sarcopenia. This method is based on previous scientific research and is aimed at minimizing pharmacotherapy. The aim is to combat symptoms and complaints and to stop (preventive) medication as much as possible
  Arms: deprescribing pharmacotherapy approach (DPA)
Other: STOPP-START deprescribing approach (SSA) — The usual care in the geriatric medicine in the Netherlands consisting of a medication review based on the STOPP-START criteria. These criteria have been combined in a protocol that describes when certain medication(groups) must be continued or discontinued for specific patient characteristics.
  Arms: STOPP-START deprescribing approach (SSA)

SUMMARY:
The goal of this clinical trial is to compare the effects of a deprescribing pharmacotherapy approach to the STOPP-START approach (usual care) in geriatric patients with sarcopenia and polypharmacy. The main question it aims to answer is the number and type of medication that can be stopped in this population without being restarted within 6 months.

After inclusion a medication review is performed by a team consisting of the researcher, a geriatrician and a hospital pharmacist, according to the protocol within which the patient was randomised. Participants are follow up at appointments after 1, 3 and 6 months. At these appointments, questionnaires are administered about the quality of life and complications related to medication.

DETAILED DESCRIPTION:
Rationale Acutely ill hospitalized geriatric patients have co-morbid disease and polypharmacy and 2/3 have low muscle strength and low muscle mass, called sarcopenic. Although all efforts are done by the multidisciplinary team to combat health problems and negative sequalae of sarcopenia, 80% of the (severely) sarcopenic patients will be deceased within 2 years. Optimalization medication is part of this multidisciplinary treatment strategy. The STOPP START criteria are applied to optimize the polypharmacy. However, it is not known whether this strategy actually results in a better or worse outcome for these patients. The question that arises is whether it is even better to minimize pharmacotherapy in these patients and only apply it if the aim is to combat symptoms and complaints and to stop (preventive) medication as much as possible. The latter is called a deprescribing pharmacotherapy approach (DPA) and seemed to be successful in a previous study concerning older frail patients.

Objective:

The effects of DPA compared to STOPP-START approach (SSA) prescribing on adverse drug reactions, medical complications, hospital readmission, quality of life in hospitalized geriatric patients with sarcopenia

Study design:

Prospective randomised intervention study. Patients will be randomised in two groups: intervention group (IG) with a DPA of 80 patients and an control group (CG) of 80 patients with a SSA.

Study population:

Acutely ill geriatric patients with sarcopenia and polypharmacy admitted to the acute care geriatric ward of Zuyderland Medical Centre.

Intervention:

Medication review in patients randomised to the IG group will be performed according to the principles of DPA and in the CG this will be performed following the SSA approach.

Main study parameters/endpoints:

Primary endpoint: the number and type of medication stopped and not restarted during medication review and number and type of medication restarted within 1, 3 and 6 months. Secondary endpoints: number and severity of Adverse Drug Reactions (ADR) and complications due to medication (e.g. delirium or falls), hospital readmission, quality of life (QoL) and mortality

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

In either of the two strategies of reviewing medication (SSA or DPA) there are risks for the sarcopenic patients with polypharmacy as part of the usual care. Applying the SSA, which is actually the usual care in the Dutch geriatric ward, there is serious risk of overtreatment with a risk of ADR and complications with holding off benefit because of a necessary time until benefit compared to the limited life expectancy. Although the risk for a ADR is low, a ADR with different kinds of impact can be expected however when starting e.g. preventive medication. But withholding preventative medication as part of DPA can cause a new health problem with minor to major impact if the life expectancy seems longer than predicted and exceeds the time until benefit. Overall, the aim of DPA is to optimize pharmacotherapy and reduce ADR, medication related complications and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years and older
* Being frail according the Groningen Frailty Indicator (GFI score >3)
* Severely sarcopenic according the European Working Group On Sarcopenia-2 criteria (EWGSOP-2) based on handgrip strength (men < 27kg and women < 16kg), appendicular skeletal muscle mass (men < 7,0 kg/m2 and women < 5,5 kg/m2) and physical function below cut-off values (Short Physical Performance Battery <9)
* The use of 5 or more different medications before hospitalization

Exclusion Criteria:

* Being not instructible
* Having an implantable cardioverter defibrillator (ICD)
* No informed consent can be optained with the participant or a legal representative

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-02-27 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Deprescribing | 6 months
  The number and type of medication stopped and not restarted during medication review and number and type of medication restarted within 1, 3 and 6 months

SECONDARY OUTCOMES:
Adverse Drug Reactions (ADR) | 6 months
  Number and severity of adverse drug reactions (ADR)
Complications due to medication | 6 months
  Number and severity of complications due to medication
Hospital readmission | 6 months
  Hospital readmission during follow up
The quality of life | 6 months
  Quality of life, obtained through questionnaires
Mortality | 6 months
  Mortality during follow up

IPD SHARING:
Plan to Share IPD: Undecided